CLINICAL TRIAL: NCT04576598
Title: Assessment of the Level of Physical Activity and Sedentarism of Stroke Survivors in the Valencian Community and Development of a Specific Self-management Program
Brief Title: Sedentarism of Stroke Survivors in the Valencian Community and Development of a Self-management Program
Acronym: SEDMA_Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Generalitat Valenciana (Other)
Responsible Party: Principal Investigator, M Luz Sanchez, PhD, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GV/2019/161
Record Dates: First submitted 2020-09-10; First posted 2020-10-06 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Stroke Sequelae
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-management group to increase physical activity levels (Experimental): This group will perform a self-management program along 6 months. This program will aim to increase the level of physical activity and adherence to healthier lifestyle habits and will be carried out through several sessions that will incorporate: education, goal setting, identification of barriers, self-control and feedback.
  Interventions: Other: Self-management program to increase physical activity levels
- Control group (Active Comparator): This group will participate in the initial educational session and will be given a leaflet with recommendations for physical activity to follow throughout the six months.
  Interventions: Other: Education information

INTERVENTIONS:
Other: Self-management program to increase physical activity levels — Information and Communication Technologies will be used to carry out various remote sessions. The sessions will address important issues to promote self-management of sedentary lifestyle by stroke survivors. Additionally, a peer support group will be created in order to improve adherence to the program.
  Other Names: Physiotherapy; Physical therapy; Physical exercise program
  Arms: Self-management group to increase physical activity levels
Other: Education information — Education on the importance of active lifestyle habits post-stroke.
  Arms: Control group

SUMMARY:
Stroke is the third leading cause of disability worldwide. Women present a higher incidence of this pathology and prevalence of its risk factors. Similarly, after stroke, women have a poorer functional outcome, higher rates of institutionalization and greater dependence on activities of daily living. People who have suffered a stroke are at increased risk of cardiovascular disease, with an estimated one-third of stroke survivors suffering a new event in the following 5 years. Current scientific literature recommends the promotion of physical activity (PA) and exercise for the prevention of stroke and its sequelae. However, stroke survivors are often insufficiently active. Therefore, changing their behavior with respect to PA and sedentary lifestyle is fundamental. Moreover, gender perspective, should also taken into account.

Thus, our aims are to study whether there are differences in women with chronic stroke sequelae compared to men in: 1) the amount of sitting time and its context, as well as the time spent in different intensities of PA; 2) the reduction of sitting time and its effect on health after the completion of the PA self-management program and sedentary lifestyle developed in this project; 3) the presence of sarcopenia, osteoporosis and the state of frailty.

To achieve these objectives, the lifestyle habits of 128 subjects (64 women) who live in the community and have chronic sequelae of stroke (≥ 6 months) will be evaluated. In addition, possible differences in the study variables will be verified with control people without sequelae of stroke. Moreover, in order to reduce the risks of stroke survivors, a program of self-management of PA and sedentary lifestyle will be developed. This program will be carried out through several sessions spread over six months that will incorporate: education, goal setting, identification of barriers, self-control and feedback. The feasibility of this intervention will be determined by examining compliance, duration, utility, and safety. At least 64 of the previously studied subjects will participate in this program, analyzing whether it favors the reduction of sitting time and its effect on health thanks to the measurement of different physical capacities. The differences between men and women in response to the program will be determined. Finally, we will explore whether the effect of the program is greater when it is implemented in the subacute than in the chronic phase.

ELIGIBILITY:
Inclusion Criteria:

* having sequelae after stroke of at least 6 months of evolution
* being community-dwelling (minimum 2 months since the last stroke)
* having the ability to walk around the house with or without technical aids but without requiring supervision from another person (FACHS ≥ 2)
* having enough cognitive capacity to provide informed consent and to understand and answer the questions proposed

Exclusion Criteria:

* not having a strength deficit in the lower limbs or walking difficulties
* having poor vital prognosis or suffering from other pathologies or disorders that may alter the development of the study (blindness, severe sensitivity alteration, musculoskeletal or cardiovascular conditions that contraindicate the performance of physical activity...)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Physical activity level at a year | 1 year
  International Physical Activity Questionnaire (IPAQ)
Change from Baseline Sedentary time at a year | 1 year
  ActiGraph wGT3X-BT accelerometers

SECONDARY OUTCOMES:
Change from Baseline Functional Mobility at a year | 1 year
  Timed Up and Go Test
Change from Baseline Lower extremity functioning at a year | 1 year
  Short Physical Performance Battery (SPPB)
Change from Baseline Postural stability in standing at a year | 1 year
  Posturography with the Wii Balance Board
Change from Baseline Frailty at a year | 1 year
  Fried's frailty phenotype
Change from Baseline Sarcopenia at a year | 1 year
  Bioimpedance with Tanita BC-418MA
Change from Baseline Bone mineral density at a year | 1 year
  Ultrasound bone densitometry with Sonost3000
Change from Baseline Motion analysis at a year | 1 year
  Inertial sensors based motion capture system Xsens-DOT

CONTACTS AND LOCATIONS:
Overall Officials: M.Luz Sánchez Sánchez, PhD, Principal Investigator — University of Valencia
Locations (2):
- Spain (2):
  - Department of Physiotherapy. University of Valencia, Valencia
  - University of Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Veerbeek JM, van Wegen E, van Peppen R, van der Wees PJ, Hendriks E, Rietberg M, Kwakkel G. What is the evidence for physical therapy poststroke? A systematic review and meta-analysis. PLoS One. 2014 Feb 4;9(2):e87987. doi: 10.1371/journal.pone.0087987. eCollection 2014. PMID 24505342
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Blaha MJ, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Judd SE, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Mackey RH, Magid DJ, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Mussolino ME, Neumar RW, Nichol G, Pandey DK, Paynter NP, Reeves MJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2014 update: a report from the American Heart Association. Circulation. 2014 Jan 21;129(3):e28-e292. doi: 10.1161/01.cir.0000441139.02102.80. Epub 2013 Dec 18. No abstract available. PMID 24352519
- [Background] Lynch EA, Jones TM, Simpson DB, Fini NA, Kuys SS, Borschmann K, Kramer S, Johnson L, Callisaya ML, Mahendran N, Janssen H, English C; ACTIOnS Collaboration. Activity monitors for increasing physical activity in adult stroke survivors. Cochrane Database Syst Rev. 2018 Jul 27;7(7):CD012543. doi: 10.1002/14651858.CD012543.pub2. PMID 30051462
- [Background] Howe MD, McCullough LD. Prevention and management of stroke in women. Expert Rev Cardiovasc Ther. 2015 Apr;13(4):403-15. doi: 10.1586/14779072.2015.1020300. Epub 2015 Mar 6. PMID 25747877
- [Background] Bushnell CD, Reeves MJ, Zhao X, Pan W, Prvu-Bettger J, Zimmer L, Olson D, Peterson E. Sex differences in quality of life after ischemic stroke. Neurology. 2014 Mar 18;82(11):922-31. doi: 10.1212/WNL.0000000000000208. Epub 2014 Feb 7. PMID 24510493
- [Background] Mackie P, Weerasekara I, Crowfoot G, Janssen H, Holliday E, Dunstan D, English C. What is the effect of interrupting prolonged sitting with frequent bouts of physical activity or standing on first or recurrent stroke risk factors? A scoping review. PLoS One. 2019 Jun 13;14(6):e0217981. doi: 10.1371/journal.pone.0217981. eCollection 2019. PMID 31194799
- [Background] Gordon NF, Gulanick M, Costa F, Fletcher G, Franklin BA, Roth EJ, Shephard T; American Heart Association Council on Clinical Cardiology, Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention; the Council on Cardiovascular Nursing; the Council on Nutrition, Physical Activity, and Metabolism; and the Stroke Council. Physical activity and exercise recommendations for stroke survivors: an American Heart Association scientific statement from the Council on Clinical Cardiology, Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention; the Council on Cardiovascular Nursing; the Council on Nutrition, Physical Activity, and Metabolism; and the Stroke Council. Stroke. 2004 May;35(5):1230-40. doi: 10.1161/01.STR.0000127303.19261.19. No abstract available. PMID 15105522
- [Background] Prior PL, Suskin N. Exercise for stroke prevention. Stroke Vasc Neurol. 2018 Jun 26;3(2):59-68. doi: 10.1136/svn-2018-000155. eCollection 2018 Jun. PMID 30191075
- [Background] Jones F, Riazi A. Self-efficacy and self-management after stroke: a systematic review. Disabil Rehabil. 2011;33(10):797-810. doi: 10.3109/09638288.2010.511415. Epub 2010 Aug 27. PMID 20795919
- [Background] Preston E, Dean CM, Ada L, Stanton R, Brauer S, Kuys S, Waddington G. Promoting physical activity after stroke via self-management: a feasibility study. Top Stroke Rehabil. 2017 Jul;24(5):353-360. doi: 10.1080/10749357.2017.1304876. Epub 2017 Mar 23. PMID 28335690